CLINICAL TRIAL: NCT05425563
Title: Effects of Expectations on Negative Affect, Perceived Cognitive Effort, and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tor Wager, Principal Investigator, Trustees of Dartmouth College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00031937; 5R01MH076136 (NIH)
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Placebo; Expectations
Keywords: Social Placebo; Somatic Pain; Vicarious Pain; Cognitive Effort
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Intervention Model Description: Within-participant design with behavioral manipulations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cue-established expectations (Experimental): Prior to experiencing the stimuli from three tasks (somatic pain/cognitive effort/vicarious pain), the participant is presented with an expectancy cue. The cue depicts 10 data points on a semi-circular scale (0-180 degrees) with categorical labels ranging from "no effort" to "strongest effort of any kind." Subsequently, participants report expectation ratings and outcome ratings.
  Interventions: Behavioral: Pain Expectancy Cues; Behavioral: Vicarious Pain Expectancy Cues; Behavioral: Cognitive Effort Expectancy Cues

INTERVENTIONS:
Behavioral: Pain Expectancy Cues — Participants are presented with a social cue that represents how previous participants responded to the upcoming somatic pain stimulus. In actuality, the cue is a social placebo, constructed by the experimenters and varying in intensity.
Behavioral: Vicarious Pain Expectancy Cues — Participants are presented with a social cue that represents how previous participants responded to the upcoming vicarious pain stimulus. In actuality, the cue is a social placebo, constructed by the experimenters and varying in intensity.
Behavioral: Cognitive Effort Expectancy Cues — Participants are presented with a social cue that represents how previous participants responded to the upcoming cognitive effort stimulus. In actuality, the cue is a social placebo, constructed by the experimenters and varying in intensity.

SUMMARY:
The investigators administer a functional neuroimaging task to investigate the effect of cue expectancy on participants' self-reported ratings across a variety of affective and cognitive domains. The experiment incorporates three tasks in which participants experience and rate 1) somatic pain, 2) vicarious pain, and 3) cognitive effort. In the somatic pain task, participants receive a brief thermal stimulus administered to a site on their arm; in the vicarious pain task, participants watch a short video clip of a patient with back/shoulder pain; in the cognitive effort task, participants perform a cognitively demanding "mental rotation" task that requires them to indicate whether two 3D objects are the same or different when rotated along the y-axis. Each trial follows a sequence that begins with a fixation, followed by a social influence cue, then an expectation rating, followed by a condition-specific stimulus, and then, an actual rating of the outcome experience.

There are four events of interest: 1) cue perception, 2) expectation rating, 3) stimulus experience, and 4) outcome rating.

First, participants are presented with a cue that depicts how other participants responded to the upcoming stimulus ("cue perception"). Although the participant is told these are real ratings, they are in fact, fabricated data points that vary in intensity (low, high). Then, based on the provided cues, participants are prompted to report their expectation of the upcoming stimulus intensity ("expectation rating") After providing an expectation rating, participants are presented with a condition-specific stimulus (somatic pain, vicarious pain, or cognitive effort) that also varies in three levels of low, medium, high stimulus intensity ("stimulus experience"). Once the stimulus presentation has concluded, participants are prompted to provide an actual rating of their experience ("outcome rating"). For the somatic pain condition, participants rate their expectations and actual experience of how painful the stimulus was; for the vicarious pain condition, they rate their expectations and actual perception of how much pain the patient was in; and for the cognitive condition, the participant provides expectation and actual ratings of task difficulty.

ELIGIBILITY:
Inclusion Criteria:

* Capable of performing experimental tasks (e.g., are able to read, can tolerate the maximum level of thermal pain stimuli).
* Fluent or native speakers of English

Exclusion Criteria:

* Contraindications to magnetic resonance scanning (e.g., metal in body, claustrophobia, pregnancy)
* Substance abuse within the last six months
* Current or recent history of pathological pain
* Current or recent history of neurological disorders
* Currently or recent history of chronic pain
* Left-handed only

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tor D Wager, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators are strongly committed to contributing to open and reproducible science. De-identified data will be shared via public online platforms such as the Open Science Framework (OSF), OpenFMRI, OpenNeuro, NeuroVault, and/or the National Institute of Mental Health Data Archive (NDA). All scripts developed to analyze data for this project will be made publicly available on Github (https://github.com/canlab/CanlabCore) at the time of publication of primary manuscripts.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: All data will be de-identified prior to sharing. Raw data will be submitted to the NDA in accordance with the terms and conditions outlined on their website (https://ndar.nih.gov/contribute_data_sharing_regimen.html) and will be publicly released within one year from the end of data collection or 6 months from the acceptance date of the first primary study manuscript on the full dataset (excluding methods development papers), whichever is later. Analyzed data/maps of statistical results and models accompanying each paper will be submitted to public repositories (OSF, OpenFMRI, OpenNeuro, and/or NeuroVault) when the primary study manuscript is accepted. All data will be shared indefinitely.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cue-established Expectations: Participants view a cue that informs them of an upcoming stimulus intensity. The purpose is to identify whether different cue levels modulate stimulus experience across somatic pain, vicarious pain, and cognitive effort domains.
Period: Overall Study
Arm/Group | Cue-established Expectations
Started | 133
Completed | 116
Not Completed | 17
Not completed — Withdrawal by Subject | 17

BASELINE CHARACTERISTICS:
Arm/Group | Cue-established Expectations
Number analyzed (Participants) | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 116
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.72 (5.52)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Male | 45
  Sex/Gender: Female | 69
  Sex/Gender: Other | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 97
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 86
  More than one race | 7
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 116

OUTCOME MEASURES:

1. Primary Outcome: Behavioral: Within Participant Subjective Outcome Ratings of Acute Thermal Pain Following High Compared to Low Cues
Description: The outcome measure is the "subjective outcome rating" for perceived pain. In each session, participants undergo pain tasks with multiple thermal stimuli. After each stimulus, participants rate their perceived pain on a semi-circular scale (0-180°). Higher angles indicate greater perceived pain. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average rating after high cue and after low cue. The final outcome is the difference between these averages, forming a contrast score that reflects the average difference in perceived pain as a function of high and low cue exposure.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened pain perception.
Time Frame: Within trials, outcome ratings are collected post-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, and contrasted to a single outcome measure: perceived pain as a function of high low cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Pain Task; Cue-modulated Stimulus Intensity: Participants view a cue that informs them of an upcoming stimulus intensity. The purpose is to identify whether different cue levels modulate stimulus experience across somatic pain, vicarious pain, and cognitive effort domains.
Arm/Group | Pain Task; Cue-modulated Stimulus Intensity
Number analyzed (Participants) | 116
units on a scale | 8.20 (0.89)
Statistical Analysis 1: Comparison: Pain Task; Cue-modulated Stimulus Intensity; Test type: Other; p < .001, Mixed Models Analysis; Slope = 8.3269, Standard Error of Mean 0.8792

2. Primary Outcome: Behavioral: Within Participant Subjective Outcome Ratings of Vicarious Pain Following High Compared to Low Cues
Description: The outcome measure is the "subjective outcome rating" for perceived vicarious pain. In each session, participants undergo vicarious pain tasks, watching multiple videos of patients in pain. After each stimulus, participants rate their perceived vicarious pain on a semi-circular scale (0-180°). Higher angles indicate that participants perceived greater pain for the patient in video. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average outcome rating after high cue and after low cue. The final outcome is the difference between these averages, forming a contrast score that reflects the average difference in perceived vicarious pain as a function of high and low cue exposure.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened perception of vicarious pain.
Time Frame: Within trials, outcome ratings are collected post-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, and contrasted to a single outcome measure: perceived vicarious pain as a function of high low cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Vicarious Pain Task; Cue-modulated Stimulus Intensity: Participants view a cue that informs them of an upcoming stimulus intensity. The purpose is to identify whether different cue levels modulate stimulus experience across somatic pain, vicarious pain, and cognitive effort domains.
Arm/Group | Vicarious Pain Task; Cue-modulated Stimulus Intensity
Number analyzed (Participants) | 116
units on a scale | 7.72 (0.66)
Statistical Analysis 1: Comparison: Vicarious Pain Task; Cue-modulated Stimulus Intensity; Test type: Other; p < .001, Mixed Models Analysis; Slope = 8.0809, Standard Error of Mean 0.5414

3. Primary Outcome: Behavioral: Within Participant Subjective Ratings of Cognitive Effort Following High Compared to Low Cues
Description: The outcome measure is the "subjective outcome rating" for cognitive effort. In each session, participants undergo cognitive effort task where images of mentally rotated figures are presented. After each stimulus, participants rate their perceived cognitive effort on a semi-circular scale (0-180°). Higher angles indicate greater perceived of cognitive effort. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average outcome rating after high cue and after low cue. The final outcome is the difference between these averages, forming a contrast score that reflects the average difference in perceived cognitive effort as a function of high and low cue exposure.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened perception of cognitive effort..
Time Frame: Within trials, outcome ratings are collected post-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, and contrasted to a single outcome measure: perceived cognitive effort as a function of high low cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Cognitive Effort Task; Cue-modulated Stimulus Intensity: Prior to experiencing the stimuli from three tasks (somatic pain/cognitive effort/vicarious pain), the participant is presented with an expectancy cue. The cue depicts 10 data points on a semi-circular scale (0-180 degrees) with categorical labels ranging from "no effort" to "strongest effort of any kind." Subsequently, participants report expectation ratings and outcome ratings.
  Pain Expectancy Cues: Participants are presented with a social cue that represents how previous participants responded to the upcoming somatic pain stimulus. In actuality, the cue is a social placebo, constructed by the experimenters and varying in intensity.
  Vicarious Pain Expectancy Cues: Participants are presented with a social cue that represents how previous participants responded to the upcoming vicarious pain stimulus. In actuality, the cue is a social placebo, constructed by the experimenters and varying in intensity.
  Cognitive Effort Expectancy Cues: Participants are presented with a social cue that represents how previous participants responded to the upcoming cognitive effort stimulus. In actuality, the cue is a social placebo, constructed by the experimenters and varying in intensity.
Arm/Group | Cognitive Effort Task; Cue-modulated Stimulus Intensity
Number analyzed (Participants) | 116
units on a scale | 8.02 (0.70)
Statistical Analysis 1: Comparison: Cognitive Effort Task; Cue-modulated Stimulus Intensity; Test type: Other; p < .001, Mixed Models Analysis; Slope = 8.121, Standard Error of Mean 0.481

4. Primary Outcome: Behavioral: Within Participant Subjective Outcome Ratings of Acute Thermal Pain Following High Cues
Description: This outcome measure is the least metabolized data of "subjective outcome rating" for perceived pain. In each session, participants undergo pain tasks with multiple thermal stimuli. After each stimulus, participants rate their perceived pain on a semi-circular scale (0-180°). Higher angles indicate greater perceived pain. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average rating after high cue and after low cue. Reported here is the average subjective outcome rating, post-high cue.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened pain perception.
Time Frame: Within trials, outcome ratings are collected post-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, reflecting: perceived pain as a function of high cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pain Task; Cue-modulated Stimulus Intensity
Number analyzed (Participants) | 116
units on a scale | 70.22 (2.85)

5. Primary Outcome: Behavioral: Within Participant Subjective Outcome Ratings of Acute Thermal Pain Following Low Cues
Description: This outcome measure is the least metabolized data of "subjective outcome rating" for perceived pain. In each session, participants undergo pain tasks with multiple thermal stimuli. After each stimulus, participants rate their perceived pain on a semi-circular scale (0-180°). Higher angles indicate greater perceived pain. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average rating after high cue and after low cue. Reported here is the average subjective outcome rating post-low cue.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened pain perception.
Time Frame: Within trials, outcome ratings are collected post-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, reflecting: perceived pain as a function of low cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pain Task; Cue-modulated Stimulus Intensity
Number analyzed (Participants) | 116
units on a scale | 61.69 (2.86)

6. Primary Outcome: Behavioral: Within Participant Subjective Outcome Ratings of Vicarious Pain Following High Cues
Description: The outcome measure is the least metabolized data of "subjective outcome rating" for perceived vicarious pain. In each session, participants undergo vicarious pain tasks, watching multiple videos of patients in pain. After each stimulus, participants rate their perceived vicarious pain on a semi-circular scale (0-180°). Higher angles indicate that participants perceived greater pain for the patient in video. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average outcome rating after high cue and after low cue. Reported here is the average subjective outcome rating post high cue.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened perception of vicarious pain.
Time Frame: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vicarious Pain Task; Cue-modulated Stimulus Intensity
Number analyzed (Participants) | 116
units on a scale | 30.66 (1.21)

7. Primary Outcome: Behavioral: Within Participant Subjective Outcome Ratings of Vicarious Pain Following Low Cues
Description: The outcome measure is the least metabolized data of "subjective outcome rating" for perceived vicarious pain. In each session, participants undergo vicarious pain tasks, watching multiple videos of patients in pain. After each stimulus, participants rate their perceived vicarious pain on a semi-circular scale (0-180°). Higher angles indicate that participants perceived greater pain for the patient in video. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average outcome rating after high cue and after low cue. Reported here is the average subjective outcome rating post low cue.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened perception of vicarious pain.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vicarious Pain Task; Cue-modulated Stimulus Intensity
Number analyzed (Participants) | 116
units on a scale | 22.78 (1.04)

8. Primary Outcome: Behavioral: Within Participant Subjective Ratings of Cognitive Effort Following High Cues
Description: The outcome measure is the least metabolized data of "subjective outcome rating" for cognitive effort. In each session, participants undergo cognitive effort task where images of mentally rotated figures are presented. After each stimulus, participants rate their perceived cognitive effort on a semi-circular scale (0-180°). Higher angles indicate greater perceived of cognitive effort. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average outcome rating after high cue and after low cue. Reported here is the average subjective outcome rating post high cue.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened perception of cognitive effort.
Time Frame: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Cognitive Effort Task; Cue-modulated Stimulus Intensity: Participants view a cue that informs them of an upcoming stimulus intensity. The purpose is to identify whether different cue levels modulate stimulus experience across somatic pain, vicarious pain, and cognitive effort domains.
Arm/Group | Cognitive Effort Task; Cue-modulated Stimulus Intensity
Number analyzed (Participants) | 116
units on a scale | 32.35 (1.38)

9. Primary Outcome: Behavioral: Within Participant Subjective Ratings of Cognitive Effort Following Low Cues
Description: The outcome measure is the least metabolized data of "subjective outcome rating" for cognitive effort. In each session, participants undergo cognitive effort task where images of mentally rotated figures are presented. After each stimulus, participants rate their perceived cognitive effort on a semi-circular scale (0-180°). Higher angles indicate greater perceived of cognitive effort. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average outcome rating after high cue and after low cue. Reported here is the average subjective outcome rating post low cue.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened perception of cognitive effort.
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Effort Task; Cue-modulated Stimulus Intensity
Number analyzed (Participants) | 116
units on a scale | 24.31 (1.19)

10. Secondary Outcome: Behavioral: Within Participant Expectation Ratings of Acute Thermal Pain Following High Compared to Low Cues
Description: The outcome measure is the "expectation rating" for upcoming pain. In each session, participants undergo pain tasks with multiple thermal stimuli. Before each stimulus, participants see a high or low cue and rate their pain expectation on a semi-circular scale (0-180°). Higher angles indicate greater pain expectations. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average rating after high cue and after low cue. The final outcome is the difference between these averages, forming a contrast score that reflects the variance in pain expectations between cues.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened expectations for thermal pain intensity.
Time Frame: Within trials, outcome ratings are collected post-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, and contrasted to a single outcome measure: expectations of pain as a function of high low cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Pain Task; Cue-established Expectations: Participants view a cue that informs them of an upcoming stimulus intensity. The purpose is to identify whether different cue levels modulate stimulus experience across somatic pain, vicarious pain, and cognitive effort domains.
Arm/Group | Pain Task; Cue-established Expectations
Number analyzed (Participants) | 116
units on a scale | 35.06 (1.99)
Statistical Analysis 1: Comparison: Pain Task; Cue-established Expectations; Test type: Other; p < .001, Mixed Models Analysis; Slope = 34.613, Standard Error of Mean 0.602

11. Secondary Outcome: Behavioral: Within Participant Expectation Ratings of Vicarious Pain Following High Compared to Low Cues
Description: The outcome measure is the "expectation rating" for upcoming vicarious pain. In each session, participants undergo vicarious pain tasks, watching multiple videos of patients in pain. Prior to each stimulus, participants see a high or low cue and rate their expectation of perceived vicarious pain for an upcoming stimulus experience on a semi-circular scale (0-180°). Higher angles suggest participants anticipate viewing videos of patients experiencing greater pain. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average expectation rating after high cue and after low cue. The final outcome is the difference between these averages, forming a contrast score that reflects difference in vicarious pain expectations between cues.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened expectations for vicarious pain intensity.
Time Frame: Within trials, outcome ratings are collected post-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, and contrasted to a single outcome measure: expectations of vicarious pain as a function of high low cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Vicarious Pain Task; Cue-modulated Expectations: Participants view a cue that informs them of an upcoming stimulus intensity. The purpose is to identify whether different cue levels modulate expectations for an upcoming stimulus experience
Arm/Group | Vicarious Pain Task; Cue-modulated Expectations
Number analyzed (Participants) | 116
units on a scale | 33.02 (1.52)
Statistical Analysis 1: Comparison: Vicarious Pain Task; Cue-modulated Expectations; Test type: Other; p = .001, Mixed Models Analysis; Slope = 33.9754, Standard Error of Mean 0.426

12. Secondary Outcome: Behavioral: Within Participant Expectation Ratings of Cognitive Effort Following High Compared to Low Cues
Description: The outcome measure is the "expectation rating" for upcoming cognitive effort. In each session, participants undergo cognitive effort tasks where images of mentally rotated figures are presented. Before each stimulus, participants see a high or low cue and rate their expectations on cognitive effort on a semi-circular scale (0-180°). Higher angles indicate greater expectations of cognitive effort. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average expectation rating after high cue and after low cue. The final outcome is the difference between these averages, forming a contrast score that reflects the difference in cognitive effort expectations between cues.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened expectations of cognitive effort.
Time Frame: Within trials, outcome ratings are collected post-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, and contrasted to a single outcome measure: expectations of cognitive effort as a function of high low cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Cognitive Effort Task; Cue-established Expectations: Participants view a cue that informs them of an upcoming stimulus intensity. The purpose is to identify whether different cue levels modulate stimulus experience across somatic pain, vicarious pain, and cognitive effort domains.
Arm/Group | Cognitive Effort Task; Cue-established Expectations
Number analyzed (Participants) | 116
units on a scale | 30.76 (1.53)
Statistical Analysis 1: Comparison: Cognitive Effort Task; Cue-established Expectations; Test type: Other; p < .001, Mixed Models Analysis; Slope = 31.63, Standard Error of Mean 0.422

13. Secondary Outcome: Behavioral: Within Participant Expectations Ratings of Acute Thermal Pain Following High Cues
Description: The outcome measure is the least metabolized data of "expectation rating" for upcoming pain. In each session, participants undergo pain tasks with multiple thermal stimuli. Before each stimulus, participants see a high or low cue and rate their pain expectation on a semi-circular scale (0-180°). Higher angles indicate greater pain expectations. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average rating after high cue and after low cue. Reported here is the average expectation rating, post-high cue.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened expectations for thermal pain intensity.
Time Frame: Within trials, outcome ratings are collected pre-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, and contrasted to a single outcome measure: expectations of pain as a function of high cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pain Task; Cue-established Expectations
Number analyzed (Participants) | 116
units on a scale | 79.46 (2.86)

14. Secondary Outcome: Behavioral: Within Participant Expectations Ratings of Acute Thermal Pain Following Low Cues
Description: The outcome measure is the least metabolized data of "expectation rating" for upcoming pain. In each session, participants undergo pain tasks with multiple thermal stimuli. Before each stimulus, participants see a high or low cue and rate their pain expectation on a semi-circular scale (0-180°). Higher angles indicate greater pain expectations. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average rating after high cue and after low cue. Reported here is the average expectation rating, post-low cue.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened expectations for thermal pain intensity.
Time Frame: Within trials, outcome ratings are collected pre-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, and contrasted to a single outcome measure: expectations of pain as a function of low cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pain Task; Cue-established Expectations
Number analyzed (Participants) | 116
units on a scale | 44.65 (3.02)

15. Secondary Outcome: Behavioral: Within Participant Expectation Ratings of Vicarious Pain Following High Cues
Description: The outcome measure is the least metabolized data of "expectation rating" for upcoming vicarious pain. In each session, participants undergo vicarious pain tasks, watching multiple videos of patients in pain. Prior to each stimulus, participants see a high or low cue and rate their expectation of perceived vicarious pain for an upcoming stimulus experience on a semi-circular scale (0-180°). Higher angles suggest participants anticipate viewing videos of patients experiencing greater pain. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average expectation rating after high cue and after low cue. Reported here is the average expectation rating, post-high cue.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened expectations for vicarious pain intensity.
Time Frame: Within trials, outcome ratings are collected pre-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, reflecting perceived vicarious pain as a function of high cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vicarious Pain Task; Cue-modulated Expectations
Number analyzed (Participants) | 116
units on a scale | 48.21 (1.56)

16. Secondary Outcome: Behavioral: Within Participant Expectation Ratings of Vicarious Pain Following Low Cues
Description: The outcome measure is the least metabolized data of "expectation rating" for upcoming vicarious pain. In each session, participants undergo vicarious pain tasks, watching multiple videos of patients in pain. Prior to each stimulus, participants see a high or low cue and rate their expectation of perceived vicarious pain for an upcoming stimulus experience on a semi-circular scale (0-180°). Higher angles suggest participants anticipate viewing videos of patients experiencing greater pain. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average expectation rating after high cue and after low cue. Reported here is the average expectation rating, post-low cue.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened expectations for vicarious pain intensity.
Time Frame: Within trials, outcome ratings are collected pre-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, reflecting perceived vicarious pain as a function of low cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vicarious Pain Task; Cue-modulated Expectations
Number analyzed (Participants) | 116
units on a scale | 14.96 (1.01)

17. Secondary Outcome: Behavioral: Within Participant Expectation Ratings of Cognitive Effort Following High Cues
Description: The outcome measure is the least metabolized data of "expectation rating" for upcoming cognitive effort. In each session, participants undergo cognitive effort tasks where images of mentally rotated figures are presented. Before each stimulus, participants see a high or low cue and rate their expectations on cognitive effort on a semi-circular scale (0-180°). Higher angles indicate greater expectations of cognitive effort. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average expectation rating after high cue and after low cue. Reported here is the average expectation rating, post-high cue.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened expectations for cognitive effort.
Time Frame: Within trials, outcome ratings are collected pre-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, reflecting: perceived pain as a function of high cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Effort Task; Cue-established Expectations
Number analyzed (Participants) | 116
units on a scale | 49.39 (1.74)

18. Secondary Outcome: Behavioral: Within Participant Expectation Ratings of Cognitive Effort Following Low Cues
Description: The outcome measure is the least metabolized data of "expectation rating" for upcoming cognitive effort. In each session, participants undergo cognitive effort tasks where images of mentally rotated figures are presented. Before each stimulus, participants see a high or low cue and rate their expectations on cognitive effort on a semi-circular scale (0-180°). Higher angles indicate greater expectations of cognitive effort. The "Outcome Measure Calculation": Ratings are grouped by cue type: High or Low. Data points in each group are averaged across sessions, yielding two measures: average expectation rating after high cue and after low cue. Reported here is the average expectation rating, post-low cue.
  * Scale: 0-180°
  * Min value: 0
  * Max value: 180
  * Higher scores indicate heightened expectations for cognitive effort.
Time Frame: Within trials, outcome ratings are collected pre-stimulus (4s window); Trials are collected across 3 sessions. Ratings are then averaged, reflecting: perceived pain as a function of low cue exposure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Effort Task; Cue-established Expectations
Number analyzed (Participants) | 116
units on a scale | 18.60 (1.21)

19. Secondary Outcome: Physiological: Within Participant Changes in Skin Conductance Response Measured With a Physiological Data Acquisition Device
Description: Each session of the experiment includes somatic pain, vicarious pain, cognitive effort tasks, in which multiple stimuli are delivered. Skin conductance response will be measured continuously, using a physiological data acquisition device, "Biopac MP150". The investigators will compare the skin conductance rate in response to stimuli delivery as a function high vs. low cue presentation.
Time Frame: Measured continuously during each task, concurrent with stimulus delivery. Each task is distributed across 3 sessions. Within each task, we plan to average skin conductance rate across sessions.
Reporting Status: Not Posted

20. Secondary Outcome: Physiological: Within Participant Changes in Skin Conductance Rate Measured With a Physiological Data Acquisition Device
Description: Each session of the experiment includes somatic pain, vicarious pain, cognitive effort tasks, in which multiple stimuli are delivered. Skin conductance rate will be measured continuously, using a physiological data acquisition device, "Biopac MP150". The investigators will compare the skin conductance rate in response to stimuli delivery as a function high vs. low cue presentation.
Time Frame: as for outcome 19
Reporting Status: Not Posted

21. Secondary Outcome: Functional Magnetic Resonance Imaging (fMRI): Within Participant Changes in Brain Signals as a Function of Stimulus Intensity
Description: After each stimulus delivery, participants are prompted to indicate outcome ratings, i.e. the intensity of their stimulus experience. Ratings are recorded on a semi-circular scale (0-180 degrees), with categorical labels indicated on the scale (e.g. "no sensation" to "strongest sensation of any kind"). The investigators will analyze stimulus brain signal as a function of high vs. med vs. low stimulus intensity. We plan to construct contrasts of stimulus brain maps based on stimulus intensity of high vs. med vs. low.
Time Frame: Measured continuously during stimulus delivery, 1 hour of functional magnetic resonance imaging scanning. Each scan is conducted across 3 sessions.
Reporting Status: Not Posted

22. Secondary Outcome: Functional Magnetic Resonance Imaging (fMRI): Within Participant Changes in Brain Signals as a Function of High vs Low Cue
Description: Investigator will model the brain event of each stimulus delivery event. From this, investigator will construct contrasts between stimulus brain maps as a function of high vs. low cue. Within each task of somatic pain, vicarious pain, and cognitive effort, we plan to both 1) average brain signals and 3) also isolate each event for further analyses.
Time Frame: as for outcome 21
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored/assessed.
Description: Adverse events were not monitored/assessed.
Arm/Group | Cue-established Expectations
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT05425563/Prot_001.pdf
  • Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT05425563/SAP_002.pdf
  • Informed Consent Form (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT05425563/ICF_003.pdf